CLINICAL TRIAL: NCT03349021
Title: The Bougiecap; a New Method for Treatment of Benign Stenosis in GI Tract
Brief Title: Bougiecap for Treatment of Benign Stenosis in GI Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Alexander Meining, Head of Endoscopy, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Esophagostenosis
Keywords: esophagus; stenosis; bougienage
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Single Group interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bougiecap (Experimental): Treatment with Bougiecap instead of Savary Bougie
  Interventions: Device: Bougiecap

INTERVENTIONS:
Device: Bougiecap — Treatment of esophagel Stenosis by Bougiecap

SUMMARY:
Feasibility testing of a cap-assisted endoscopic bougienage for benign upper GI stenosis with direct optical control.

DETAILED DESCRIPTION:
Benign stenosis in the GI tract are endoscopically treated by using Savary-Gilliard Dilators. This method, although sufficient in its interventional success, provides only haptic control and often requires wire guidance or X-ray imaging for monitoring the position of the stenosis, the dilator and the dilation process.

To guarantee the missing optical feedback and enhance the intraprocedural control a conical, clear cap was developed. This single use device is attachable to the front end of an endoscope and provides direct visual evaluation of the mucosal damage and progress of the Bougienage, making x-ray imaging obsolete while resulting in an effective dilation. For the bougienage treatment, the endoscope with the cap on top is inserted into the patient's GI tract and aimed at the stenosis. By pushing the endoscope forward the cone shaped cap expands the mucosal diameter by conversion of longitudinal to radial force vectors. Lateral and frontal openings allow suction and flush during procedure.

The clear tapering cap is now to be tested for ist technical feasibility and ability to improve patients' quality of life following treatment. Therefore a quality of life questionnaire (Swal QoL) evaluating the patients' dysphagia is done right before and two weeks after the bougienage and an effective dilation is proved by being able to pass the stenosis with the endoscope after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* benign Stenosis of the esophagus
* indication for endoscopic treamtent of stenosis

Exclusion Criteria:

* no informed consent
* malignancy based Stenosis
* no indication for endoscopic treamtent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Efficient bougienage with BougieCap | Day 0 (directly) after endoscopy
  To measure the effect of bougienage a passage with the endoscope should be possible.after Treatment with the BougieCap (5mm Endoscope, 10mm endoscope)

SECONDARY OUTCOMES:
Qol dysphagia | Day 0 before endoscopy and Day14 after treatment
  Evaluation of life Quality by a 13 questions questionnaire. Clinical symptoms of dysphagia and General Quality of life are evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, Prof., Principal Investigator — Head of Endoscopy
Locations (3):
- Germany (2):
  - Universitätklinikum Ulm, Ulm, Baden-Wurttemberg
  - Marienhospital, Essen
- Southhamptan University Hospital, Southhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter B, Schmidbaur S, Rahman I, Albers D, Schumacher B, Meining A. The BougieCap - a new method for endoscopic treatment of complex benign esophageal stenosis: results from a multicenter study. Endoscopy. 2019 Sep;51(9):866-870. doi: 10.1055/a-0959-1535. Epub 2019 Jul 23. PMID 31342473